CLINICAL TRIAL: NCT01066715
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging Study of the Safety and Efficacy of XOMA 052 in Subjects With Type 2 Diabetes Mellitus on Stable Metformin Monotherapy
Brief Title: Safety and Efficacy of XOMA 052 in Subjects With Type 2 Diabetes Mellitus on Stable Metformin Monotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X052078
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Type 2; Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- XOMA 052 (Experimental)
  Interventions: Drug: XOMA 052

INTERVENTIONS:
Drug: XOMA 052 — Sterile solution subcutaneously administered monthly for 6 months
  Arms: XOMA 052
Drug: Placebo — Sterile solution subcutaneously administered monthly for 6 months
  Arms: Placebo

SUMMARY:
The study hypothesis is that XOMA 052 improves glycemic control in subjects with Type 2 Diabetes.

Study X052078 is designed to establish efficacious dose(s) for future studies based on improvement in HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D (disease duration ≥ 6 months)
* HbA1c ≥ 6.8% and ≤ 10.0%
* Have been on a stable regimen of metformin monotherapy for at least 12 weeks prior to Day 0
* Willingness to maintain stable diet and exercise regime throughout the study
* Willingness to maintain current doses/regimens of vitamins and dietary supplements through the end of the study

Exclusion Criteria:

* Uncontrolled hypertension
* History of malignancy within 5 years
* History of allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Advanced stage heart failure (New York Heart Association [NYHA] class 3 or 4)
* Clinically significant uncontrolled arrhythmias
* History of tuberculosis
* Active leg, foot, or decubitus ulcer
* Any significant inflammatory, rheumatologic, or systemic autoimmune disease
* History of chronic infections
* History or any symptoms of a demyelinating disease
* Major surgery within 3 months
* Female subjects who are pregnant, planning to become pregnant

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline (Day 0 pre-dose) in HbA1c at Day 182 | Day 0 pre-dose and Day 182

SECONDARY OUTCOMES:
Safety assessed by pre- and post-treatment serial measurements of vital signs, clinical laboratory assessments, daily fasting blood glucose measured by the subject using a glucose monitor, and treatment-emergent adverse events. | Day 0 through Day 182
Diabetic parameters: mean change from baseline (Day 0 pre-dose) at measured time points | Day 0 pre-dose through Day 182
Inflammatory markers: mean change from baseline (Day 0 pre-dose) at measured time points | Day 0 pre-dose through Day 182
Markers of cardiovascular disease: mean change from baseline (Day 0 pre-dose) at measured time points | Day 0 pre-dose through Day 182
Serum levels of XOMA 052 (select sites only) | Day 28 pre-dose, Day 168 pre-dose, and Day 182

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - Huntsville, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Chino, California
  - Escondido, California
  - Los Angeles, California
  - Los Gatos, California
  - National City, California
  - Palm Springs, California
  - Sacramento, California
  - San Diego, California
  - Tarzana, California
  - Walunt Creek, California
  - Bradenton, Florida
  - Brooksville, Florida
  - Coral Gables, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Port Orange, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Newton, Kansas
  - Columbia, Maryland
  - Oxon Hill, Maryland
  - Edina, Minnesota
  - St Louis, Missouri
  - Butte, Montana
  - Henderson, Nevada
  - Las Vegas, Nevada
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Wilson, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Kettering, Ohio
  - Lynhurst, Ohio
  - Wadsworth, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Greer, South Carolina
  - Kingsport, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Orem, Utah
  - West Jordan, Utah
  - Burke, Virginia
  - Virginia Beach, Virginia
  - Renton, Washington